CLINICAL TRIAL: NCT03656848
Title: Comparison of Quantitative Flow Ratio Guided and Angiography Guided Percutaneous InterVention in Patients With cORonary Artery Disease (The FAVOR III China Study)
Brief Title: The FAVOR III China Study
Acronym: FAVORIII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Bo Xu, Director, Catheterization Laboratories, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FAVOR III China - 2508
Record Dates: First submitted 2018-08-31; First posted 2018-09-04 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease; Myocardial Ischaemia; Coronary Circulation; Coronary Stenosis; Percutaneous Coronary Intervention
Keywords: Quantitative Coronary Angiography; Quantitative Flow Ratio; Coronary Artery Disease; Myocardial Ischaemia; Percutaneous Coronary Intervention; Coronary Circulation
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Angiography; Coronary Angiography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a blinded clinical trial. Subjects and clinical assessor will be blinded to the assignment results. All the study site personnel will receive training for the blinding measures before the trial initiating. In addition to standard procedural sedation, music-playing headphones will be worn by the patient during the whole procedure, and patients in both groups will be preset a 10 minutes delay for QFR calculation before the PCI procedure, a lesion/device evaluation form is required to fill in during the period in both groups, to reduce the possibility of unblinding. All the study site personnel will be trained not to disclose the treatment assignment to the subject in any unplanned time. Subject blinding should be maintained until the one-year follow-up visit for all registered subjects is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QFR-guided PCI group (Experimental): If the patient is assigned to QFR-guided PCI, QFR is first measured in all coronary arteries with DS% ≥ 50% and ≤ 90%. Then PCI treatment is performed in lesions with QFR ≤ 0.80, and optimal medicine treatment is prescribed to those with QFR > 0.80. It is strongly recommended to select the device size based on the 3D-QCA measurements in this group.
  Interventions: Diagnostic Test: QFR; Diagnostic Test: Angiography
- Angiography-guided PCI group (Active Comparator): If the patient is assigned to angiography-guided PCI, then the investigator performs PCI according to the stenosis severity based on visual assessment of the angiogram. No other functional tests such as FFR/iFR can be used for further assessment of the lesion before PCI.
  Interventions: Diagnostic Test: Angiography

INTERVENTIONS:
Diagnostic Test: QFR — QFR is a novel method for evaluating the functional significance of coronary stenosis by calculation of the pressure drop in the vessel based on two angiographic projections.
  Other Names: Quantitative Flow Ratio
  Arms: QFR-guided PCI group
Diagnostic Test: Angiography — Coronary angiography is a procedure that uses contrast under x-ray pictures to detect stenosis in the coronary arteries
  Other Names: Coronary angiography

SUMMARY:
The overall purpose of the FAVOR III China trial is to investigate if a strategy of quantitative flow ratio (QFR)-guided percutaneous coronary intervention (PCI) yields superior clinical outcome and cost-effectiveness compared to a strategy of standard coronary angiography-guided PCI in evaluation of patients with coronary artery disease.

DETAILED DESCRIPTION:
The FAVOR III China is a prospective, multicenter, blinded, randomized, superiority clinical trial comparing the clinical outcome and cost-effectiveness of the two PCI strategies, QFR-augmented angiography-guided (QFR-guided) strategy versus an angiography-only-guided (angiography-guided) strategy , in evaluation of patients with coronary artery disease (CAD). The study is adequately powered to detect if the primary outcome by the QFR-guided PCI strategy is superior to the standard angiography-guided PCI strategy. The hypothesis is that a QFR-guided PCI strategy results in superior clinical outcome, assessed by rate of Major Adverse Cardiac Events (MACE) defined as a composite of all-cause mortality, any myocardial infarction (MI) and any ischemia-driven revascularization at 1 year, compared to a standard angiography-guided PCI strategy. If QFR-guided strategy is shown to be superior to the angiography-guided strategy, the lower clinical costs and better clinical outcome by QFR may suggest it to be the preferred strategy for invasive functional evaluation of coronary artery stenosis.

The primary and major secondary endpoints will be analyzed in prespecified subgroups, including age, sex, diabetes, smoking status, acute coronary syndrome, body mass index, left ventricular ejection fraction, lesion location, length and reference vessel diameter, stenosis severity, multivessel disease, calcified lesion, bifurcation, tandem and bending/tortuous lesion, QFR gray zone (0.75-0.85), QFR based functional and residual functional SYNTAX score, residual QFR, center experience for invasive physiology, and learning experience with QFR.

For the purpose of protecting trial subjects and study personnel while maintaining trial data integrity during the coronavirus disease 2019 (COVID-19) pandemic, we particularly arranged an unscheduled telephone follow-up for all the participants, to evaluate the potential impact of the pandemic. Using a special designed follow-up questionnaire, all subjects were required to report the presence of COVID-19 infection and its related complications, any possible ischemia symptom, any hospitalization or outpatient visit, and interruption of cardiovascular medicine during this time (from Jan 20, 2019 to May 1, 2020). Clinical event committees (CEC) will update the working protocol to enable the re-adjudication of events from the onset of the pandemic to the end of the trial. All the events will be classified as related, possibly related, or not related to COVID-19 infection. To identify the interaction between COVID-19 pandemic and randomized revascularization strategy in the current study, several prespecified subsets will be added to the subgroups analysis, including COVID-19 positive vs. negative subjects, pre-pandemic vs. during pandemic vs. post-pandemic subjects, and the sites located at the high-risk region vs. low- to mediate-risk region.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* Age ≥ 18 years
* Stable or unstable angina pectoris, or post-acute myocardial infarction (≥ 72 hrs)
* Signed written informed consent
* Eligible for PCI by the operators

Angiographic inclusion criteria:

* At least one lesion is present of DS% ≥50% and ≤90% in one major native epicardial coronary artery and supplying viable myocardium
* Reference lumen diameter ≥ 2.5mm by visual assessment

Exclusion Criteria:

General exclusion criteria:

* Cardiogenic shock or severe heart failure (NYHA ≥III)
* Severely impaired renal function: creatinine > 150μmol/L or Cockcroft-Gault calculated GFR < 45 ml/kg/1.73 m2
* Allergy to iodine-containing contrast agents
* Pregnancy or intention to become pregnant during the course of the trial
* Life expectancy less than one year

Angiographic exclusion criteria:

* With only one coronary artery lesion（DS%>90%）with TIMI flow < 3
* Target stenoses are culprit lesions related with acute myocardial infarction
* Target stenoses in the vessel involving myocardial bridge
* Poor angiographic image quality precluding vessel contour detection or with suboptimal contrast filling
* Severe overlap in the stenosed segment or severe tortuosity of any target vessel deemed unable for QFR measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3847 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2025-02-19 (Estimated)

PRIMARY OUTCOMES:
MACE | 1 year
  A composite of all-cause mortality, any myocardial infarction and any ischemia-driven revascularization

SECONDARY OUTCOMES:
MACE excluding peri-procedural MI (Major secondary endpoint) | 1 year
  all-cause mortality, any spontaneous myocardial infarction and any ischemia-driven revascularization
MACE | 1 month, 2 years, 3 years, 4 years and 5 years
  A composite of all-cause mortality, any myocardial infarction and any ischemia-driven
Death | 1 month, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  Cardiovascular, non-cardiovascular and undetermined death
MI | 1 month, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  Target vessel related and non-target vessel related MI
Target vessel revascularization (TVR) | 1 month, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  The ischemia driven and non-ischemia driven TVR
Any coronary artery revascularization | 1 month, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  The The ischemia driven and non-ischemia driven Revascularization
Definite or probable stent thrombosis | 1 month, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  Definite and probable stent thrombosis during acute, sub-acute, late, and very late phase according to the Academic Research Consortium (ARC)-2
The PCI strategy changes based on the QFR and 3D-QCA | During the procedure
  PCI strategy changes following QFR and three-dimension quantitative coronary angiography (3D-QCA)
Cost during 1-year follow-up | 1 month, 6 months, 1 year
  Costs include direct clinical costs during the initial hospitalization and other resources used, main cardiovascular medication expenses, and outpatient and/or hospitalization expenses associated with MACE.
Quality-adjusted-life-years (QALYs) index | 1 month, 6 months, 1 year
  QALYs determined using EuroQol five dimensions questionnaire (EQ-5D) in official Chinese version, to assess the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Xu, MBBS, Principal Investigator — Fu Wai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences; Shubin Qiao, MD, Principal Investigator — Fu Wai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences
Locations (1):
- Fu Wai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Background] Westra J, Andersen BK, Campo G, Matsuo H, Koltowski L, Eftekhari A, Liu T, Di Serafino L, Di Girolamo D, Escaned J, Nef H, Naber C, Barbierato M, Tu S, Neghabat O, Madsen M, Tebaldi M, Tanigaki T, Kochman J, Somi S, Esposito G, Mercone G, Mejia-Renteria H, Ronco F, Botker HE, Wijns W, Christiansen EH, Holm NR. Diagnostic Performance of In-Procedure Angiography-Derived Quantitative Flow Reserve Compared to Pressure-Derived Fractional Flow Reserve: The FAVOR II Europe-Japan Study. J Am Heart Assoc. 2018 Jul 6;7(14):e009603. doi: 10.1161/JAHA.118.009603. PMID 29980523
- [Background] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Song L, Tu S, Sun Z, Wang Y, Ding D, Guan C, Xie L, Escaned J, Fearon WF, Kirtane AJ, Serruys PW, Wijns W, Windecker S, Leon MB, Stone GW, Qiao S, Xu B; FAVOR III China Investigators. Quantitative flow ratio-guided strategy versus angiography-guided strategy for percutaneous coronary intervention: Rationale and design of the FAVOR III China trial. Am Heart J. 2020 May;223:72-80. doi: 10.1016/j.ahj.2020.02.015. Epub 2020 Feb 24. PMID 32179258
- [Result] Xu B, Tu S, Song L, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Yang J, Liu X, Guo L, Shen C, Zhang Y, Zhang Q, Pan H, Fu X, Liu J, Zhao Y, Escaned J, Wang Y, Fearon WF, Dou K, Kirtane AJ, Wu Y, Serruys PW, Yang W, Wijns W, Guan C, Leon MB, Qiao S, Stone GW; FAVOR III China study group. Angiographic quantitative flow ratio-guided coronary intervention (FAVOR III China): a multicentre, randomised, sham-controlled trial. Lancet. 2021 Dec 11;398(10317):2149-2159. doi: 10.1016/S0140-6736(21)02248-0. Epub 2021 Nov 4. PMID 34742368
- [Result] Jin Z, Xu B, Yang X, Jia R, Meng S, Hu H, Deng Y, Cao X, Ruan Y, Han J, Liu J, Qu X, Zhou Y, Wang J, Fu G, Yu B, Wang Y, Guan C, Song L, Tu S, Qiao S, Stone GW; FAVOR III China Study Group. Coronary Intervention Guided by Quantitative Flow Ratio vs Angiography in Patients With or Without Diabetes. J Am Coll Cardiol. 2022 Sep 27;80(13):1254-1264. doi: 10.1016/j.jacc.2022.06.044. PMID 36137676
- [Result] Song L, Xu B, Tu S, Guan C, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Yang J, Liu X, Guo L, Shen C, Zhang Y, Zhang Q, Pan H, Zhang R, Liu J, Zhao Y, Wang Y, Dou K, Kirtane AJ, Wu Y, Wijns W, Yang W, Leon MB, Qiao S, Stone GW; FAVOR III China Study Group. 2-Year Outcomes of Angiographic Quantitative Flow Ratio-Guided Coronary Interventions. J Am Coll Cardiol. 2022 Nov 29;80(22):2089-2101. doi: 10.1016/j.jacc.2022.09.007. Epub 2022 Sep 19. PMID 36424680
- [Derived] Zhang R, Wang HY, Song L, Guan C, Yin D, Zhu C, Feng L, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Zhao Y, Wang Y, Liu W, Qiao S, Tu S, Wijns W, Dou K; FAVOR III China Study Group. Rationales Behind Physiology-Guided Revascularization: Diagnostic Impact of Quantitative Flow Ratio in the FAVOR III China Trial. JACC Cardiovasc Interv. 2025 Nov 20:S1936-8798(25)02702-5. doi: 10.1016/j.jcin.2025.10.042. Online ahead of print. PMID 41263729
- [Derived] Ding S, Zhou Z, Zou Z, Cheng F, Sheng X, Liu X, Guo L, Shen C, Zhang Y, Pan H, Xu Y, Chu M, Wang Y, Guan C, Tu S, Kirtane AJ, Qiao S, Song L, Stone GW, Pu J; FAVOR III China Study Group. Two-year outcomes of quantitative flow ratio-based physiology-guided percutaneous coronary intervention in patients with low-risk acute coronary syndrome: a prespecified secondary analysis of FAVOR III China. EClinicalMedicine. 2025 Aug 30;88:103461. doi: 10.1016/j.eclinm.2025.103461. eCollection 2025 Oct. PMID 40926902
- [Derived] Geng Y, Guan C, Jiang Y, Yang W, Yu B, Fu G, Pu J, Qu X, Zhang Q, Zhao Y, Yu L, Huang Y, Tu S, Qiao S, Song L. Prognostic impact of guideline-directed medical therapy after functionally complete revascularisation in patients with obstructive coronary artery diseases. Heart. 2025 Aug 7:heartjnl-2025-325670. doi: 10.1136/heartjnl-2025-325670. Online ahead of print. PMID 40780826
- [Derived] Dai J, Guan C, Xu X, Hou J, Jia H, Yu H, Jin Z, Fu G, Wu X, Wang L, Huang R, Shen Z, Zhao Y, Jin Y, Song L, Tu S, Qiao S, Yu B, Xu B, Stone GW; FAVOR III China study group. Angiographic Quantitative Flow Ratio-Guided Treatment of Patients With Physiologically Intermediate Coronary Lesions. J Am Heart Assoc. 2025 Apr;14(7):e035756. doi: 10.1161/JAHA.124.035756. Epub 2025 Mar 21. PMID 40118790
- [Derived] Zhao Y, Guan C, Wang Y, Jin Z, Yu B, Fu G, Chen Y, Guo L, Qu X, Zhang Y, Dou K, Wu Y, Yang W, Tu S, Escaned J, Fearon WF, Qiao S, Cohen DJ, Krumholz HM, Xu B, Song L; FAVOR III China Study Group. Cost-effectiveness of angiographic quantitative flow ratio-guided coronary intervention: A multicenter, randomized, sham-controlled trial. Chin Med J (Engl). 2025 May 20;138(10):1186-1193. doi: 10.1097/CM9.0000000000003484. Epub 2025 Mar 3. PMID 40025631
- [Derived] Chen Y, Gao L, Vogel B, Tian F, Jin Q, Guo J, Sun Z, Yang W, Jin Z, Yu B, Fu G, Pu J, Qu X, Zhang Q, Zhao Y, Yu L, Guan C, Tu S, Qiao S, Xu B, Mehran R, Song L; FAVOR III China Study Group. Sex Differences in Clinical Outcomes Associated With Quantitative Flow Ratio-Guided Percutaneous Coronary Intervention. JACC Asia. 2023 Nov 28;4(3):201-212. doi: 10.1016/j.jacasi.2023.09.012. eCollection 2024 Mar. PMID 38463683
- [Derived] Tu S, Xu B, Chen L, Hong H, Wang Z, Li C, Chu M, Song L, Guan C, Yu B, Jin Z, Fu G, Liu X, Yang J, Chen Y, Ge J, Qiao S, Wijns W; FAVOR III China Study Group. Short-Term Risk Stratification of Non-Flow-Limiting Coronary Stenosis by Angiographically Derived Radial Wall Strain. J Am Coll Cardiol. 2023 Feb 28;81(8):756-767. doi: 10.1016/j.jacc.2022.11.056. PMID 36813375